CLINICAL TRIAL: NCT04601623
Title: Ultrasound Shear Wave Elastography to Predict the Treatment Effect and Risk of Re-tear in Patients With Large-to-massive Rotator Cuff Tears
Brief Title: Ultrasound to Predict the Prognosis of Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: MOST 109-2314-B-182A-171
Record Dates: First submitted 2020-10-16; First posted 2020-10-26 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff tears; surgery; ultrasound; elastography
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sonoelastography — This diagnostic test would be executed by a physician who has experiences of using Siemens Acuson S2000 ultrasound system for more than three year. The examination includes two of four rotator cuff muscles, listed as follows, supraspinatus muscle and infraspinatus muscle. Linear transducer (4-9 MHz) would be used for the whole test. The probe would be positioned along the longitudinal axis of the muscle belly. Compressive sonoelastography technique is used for semiquantitative analysis. In order to maintain the quality of images, quality factor needs to be over or equal to 60. The quantitative analysis was performed by shear wave sonoelastography and the region of interest (ROI) would be divided into four quadrants. The physicians will measure the shear wave velocity at the center point of each quadrant.

SUMMARY:
To predict the prognosis of large-to-massive RCTs and risk of re-tear by ultrasound elastography.

DETAILED DESCRIPTION:
Most symptomatic large-to-massiverotator cuff tears (RCTs) should be operated, but the prognosis and postoperative risk of re-tear depended on the quality of rotator cuff muscles. Preoperative evaluations were usually done by magnetic resonance imaging (MRI). MRI was used in recent studies to predict the surgical outcome of large-to-massive RCTs and postoperative re-tear, but the clinical availability was not as good as ultrasound. The investigators hypothesize that ultrasound elastography can predict the prognosis of large-to-massive RCTs and risk of re-tear.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with rotator cuff tear by an orthopedist.
2. The large-to-massive rotator cuff tears need to be confirmed by magnetic resonance imaging or ultrasound. The definitions of this diagnosis include a tear over 3 cm or any full-thickness of tears in more than two rotator cuff muscles.
3. Being willing to cooperated with the arranged examinations before the operation.

Exclusion Criteria:

1. Patients who are only diagnosed with partial-thickness rotator cuff muscle tears or small- to large- sized full-thickness tears.
2. Patients who have acromioclavicular arthritis that needs distal clavicle resection.
3. Patients who had serious glenohumeral arthritis, pseudoparalysis, or any other shoulder trauma history.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator will enroll participants with diagnosis of large-to-massive rotator cuff tears who will receive surgical repairs later, and sonoelastography and MRI are necessary for preoperative evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline finding of sonoelastography | Baseline, 3 months, 6 months, 12 months
  This diagnostic test would be executed by a physician who has experiences of using Siemens Acuson S2000 ultrasound system for more than three year. The examination includes two of four rotator cuff muscles, listed as follows, supraspinatus muscle and infraspinatus muscle. Linear transducer (4-9 MHz) would be used for the whole test. The probe would be positioned along the longitudinal axis of the muscle belly. Compressive sonoelastography technique is used for semiquantitative analysis. In order to maintain the quality of images, quality factor needs to be over or equal to 60. The quantitative analysis was performed by shear wave sonoelastography and the region of interest (ROI) would be divided into four quadrants. The physicians will measure the shear wave velocity at the center point of each quadrant.

SECONDARY OUTCOMES:
Passive range of motions | Baseline, 3 months, 6 months, 12 months
  Passive range of motions of internal and external rotation, abduction, extension, and flexion, which are assessed by a goniometer.
Muscle strength | Baseline, 3 months, 6 months, 12 months
  Muscle strength assessment include the following motions, which are internal and external rotation, abduction, extension, and flexion. They are measured by a manual dynamometer
American Shoulder and Elbow Surgeons score (ASES score) | Baseline, 3 months, 6 months, 12 months
  Shoulder function is evaluated using American Shoulder and Elbow Surgeons score, which includes one item for pain (VAS) and 10 items for shoulder function. The ASES score ranges from 0 to 100, and the outcome is better when ASES score is higher.
Western Ontario Rotator Cuff Index (WORC index) | Baseline, 3 months, 6 months, 12 months
  Shoulder function is evaluated using Western Ontario Rotator Cuff Index, which includes physical symptoms (10 items), sport/recreation/work function (4 items), lifestyle function (4 items), and emotional function (3 items). The WORC index ranges from 0 to 2100 or can be converted to 0 to 100 scale, and the outcome is better when WORC index is lower.
WHOQOL-BREF (Taiwan version) | Baseline, 3 months, 6 months, 12 months
  The WHOQOL-BREF (Taiwan version) instrument comprises 28 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF (Taiwan version) is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials. The total score WHOQOL-BREF (Taiwan version) can be transformed to a 0-100 scale, and the quality of life is better when the score is higher.
EQ-5D-3L | Baseline, 3 months, 6 months, 12 months
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
MRI | Baseline, 6 months
  MRI was performed on a 1.5T system (Signa Horizon LX, GE Healthcare) equipped with a standard shoulder surface coil. The shoulder MRI protocol was identical for all patients and consisted of axial proton-density-weighted fast spinecho with fat suppression sequence, the sequences was performed above the level o f the acromioclavicular joint down to below the axillary pouch with the following parameters: Coronal oblique proton-density-weighted with and without fat suppression, with axis parallel to the supraspinatus tendon, and sagittal oblique proton-density--weighted with and without fat suppression, with axis perpendicular to the coronal oblique axis, the ast spin-echo sequences were performed with the following parameters: TR msec/TE msec, 2700-4800 /25-40, echo-train length, 6; matrix, 256 × 256; field of view, 180 mm; section thickness, 2.5 mm with 2-mm gap. No IV or intraarticular gadolinium was administered.

CONTACTS AND LOCATIONS:
Overall Officials: Po-Cheng Chen, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan